CLINICAL TRIAL: NCT01076751
Title: Observational Prospective Study of Survival, Treatment Patterns, Disease and Economic Outcomes in Patients With Metastatic Castrate-resistant Prostate Cancer (CRPC) With Progression During or After a First-line Docetaxel-based Regimen
Brief Title: Observational Registry of Treatment Patterns in Castrate-resistant Prostate Cancer (CRPC) Patients
Acronym: PORTREAT
Status: Terminated | Type: Observational
Why Stopped: delay in recruitment
Sponsor: Sanofi (Industry)
Responsible Party: Trial Transparency Team, sanofi-aventis
Other Study IDs: DIREG_C_05073
Record Dates: First submitted 2010-02-25; First posted 2010-02-26 (Estimated); Last update posted 2011-02-14 (Estimated); Status verified 2011-02

CONDITIONS: Prostatic Neoplasms
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- CRPC patients

SUMMARY:
Primary Objective:

* Describe real-life survival of CRPC patients who received first-line docetaxel and have disease progression

Secondary Objective:

* Describe treatment patterns
* Describe the characteristics and outcomes of patients who received second-line taxane-based treatment compared to others
* Describe economic and patient-reported outcomes

ELIGIBILITY:
Inclusion criteria:

* Patients with CRPC progressing during the course of first line docetaxel-based chemotherapy or after at least 3 cycles (equivalent to 225mg/m2) of first line docetaxel-based chemotherapy
* Patient who have given their written consent

Exclusion criteria:

* Current participation in a clinical trial for the second-line treatment of prostate cancer
* Patients having received less than 3 cycles of first line docetaxel-based chemotherapy and discontinued for a reason other than disease progression or toxicity
* Patients having already started a second line treatment

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with metastatic castrate-resistant prostate cancer
Sampling Method: Non-Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2010-02; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Overall survival | At Month 12 or death

SECONDARY OUTCOMES:
Sequence of treatment in second-line, third-line | At Month 6 (+/- 2 months), Month 12 or death
Characteristics and outcomes of patients who receive second-line taxane-based treatment compared to others | At baseline, Month 6 (+/- 2 months), Month 12 or death
Indicators of health care resource utilization | At baseline, Month 6 (+/- 2 months), Month 12 or death
Quality of life | At baseline, Month 6 (+/- 2 months) or Month 12

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (5):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States
- Sanofi-Aventis Administrative Office, Paris, France
- Sanofi-Aventis Administrative Office, Frankfurt, Germany
- Sanofi-Aventis Administrative Office, Barcelona, Spain
- Sanofi-Aventis Administrative Office, Guildford Surrey, United Kingdom